CLINICAL TRIAL: NCT06084832
Title: Smartphone Application for University Students With Binge Drinking Behavior: National Randomized Controlled Trial
Brief Title: Smartphone Application for University Students With Binge Drinking Behavior
Acronym: SmartBinge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: EPSM Marne, Reims (Unknown); SCA-LAB UMR-CNRS 9193, Lille (Unknown); Paul Valery University, Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PI2023_843_0069
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Drinking; Binge Drinking
Keywords: Alcohol; Binge Drinking; Phosphatidylethanol; Smartphone; Health
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Binge Drinking (Experimental)
  Interventions: Biological: blood microsampling
- Binge Drinking-control (Active Comparator)
  Interventions: Biological: blood microsampling

INTERVENTIONS:
Biological: blood microsampling — blood microsampling for the measure of Phosphatidylethanol

SUMMARY:
Alcohol use is a causal factor in more than 200 diseases and injury conditions (see ICD-10) and in France, alcohol is the first cause of hospitalization. Binge drinking (BD) has emerged as a major public health issue among student populations and is associated with negative consequences and social, cognitive and brain alterations. More than half of French university students have reported BD in the past month and are at increased risk of several alcohol-related consequences such as memory and sleep impairments, and reduced quality of life. BD is also a major risk factor in the development of alcohol addiction, with individual and environmental factors playing a role that is still poorly understood. Moreover, most students and young adults are reluctant to seek interventions when it is provided by health care professionals (only 4-5%) and have poor insight with regard to their alcohol use patterns / habits. Thus, there is an urgent need for developing effective prevention and intervention programs to reduce alcohol drinking in students. Recent studies have demonstrated that new types of technology-delivered interventions are promising tools for addressing unhealthy alcohol use. For example, an uncontrolled trial pilot study using a smartphone application-delivered intervention produced a reduction in both number of drinks per week and BD from baseline to 3-month follow-up. A recent review also showed significant outcomes of a mobile health intervention for self-control of unhealthy alcohol use. The investigators hypothesize that a timeline follow-back and personalized feedback based on the use of a mobile application can reduce excessive alcohol intake at 3-months. This study will provide scientific knowledge about BD in students, but also regarding a new type of intervention that could be effective for prevention in non-treatment seeking individuals and reducing the severity of health problems associated with excessive alcohol intake.

ELIGIBILITY:
Inclusion Criteria:

* Students between 18 and 25 years old
* AUQ score greater than or equal to 24, and AUDIT score greater than or equal to 3 for its first 3 items. Drinking details with the DDQ when necessary.
* BD behavior: at least one occasion with 6 or more drinks in the last 3 months.
* Consent to be included in the study
* Affiliated to social security

Exclusion Criteria:

* Not having a smartphone with an Apple or Android system.
* Previous use of the MyDéfi smartphone application
* Declaration of a psychiatric / neurologic condition
* Pregnant, parturient or breastfeeding woman
* Subject under guardianship, curators or restricted under public law

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 628 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change of the number of standard drinks per week | 30 months

SECONDARY OUTCOMES:
Change of the PEth concentration | 3 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 6 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 9 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 12 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 15 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 18 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 21 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 24 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 27 months
  phosphatidylethanol (PEth)
Change of the PEth concentration | 30 months
  phosphatidylethanol (PEth)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andre C, Sauton P, Dreinaza M, Diouf M, Bodeau S, Martinetti M, Trouillet R, de Groote C, Nandrino JL, Alexandre A, Benzerouk F, Gierski F, Perney P, Grellet L, Andre J, Naassila M. Effect of the MyDefi Smartphone Application on Binge Drinking Among University Students: Protocol of a Double-Blind Multicenter Prospective National Randomized Controlled Trial Using Phosphatidylethanol as a Biomarker-The SMARTBINGE Trial. Int J Methods Psychiatr Res. 2025 Jun;34(2):e70014. doi: 10.1002/mpr.70014. PMID 40165584